CLINICAL TRIAL: NCT03358420
Title: Inflammation and Steatosis: the Role of Alpha-defensin
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-103-16
Record Dates: First submitted 2017-11-27; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Inflammation; Fatty Liver
MeSH Terms: conditions — Inflammation; Fatty Liver

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Immunohistochemical staining — Pathological liver slides to be immunohistochemically stained for alpha-defensin

SUMMARY:
The aim of this study is to examine the correlation between the severity of non-alcoholic steatohepatitis/non alcoholic fatty liver disease (NASH/NAFLD) in naïve and hepatitis C (HCV) positive patients and the amplitude of alpha-defensin immunohistochemical staining in liver biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Fatty liver disease patients with liver biopsy

Exclusion Criteria:

* None

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending our liver unit who underwent a liver biopsy with proven fatty liver disease
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Amplitude of immunohistochemical stain | Six months
  The amplitude of each slide will be graded from 1-4

CONTACTS AND LOCATIONS:
Overall Officials: Rami Abu Fanne, MD, Study Director — Hillel Yaffe Medical Center
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No